CLINICAL TRIAL: NCT04756388
Title: E-SMART: Examining Strategy Monitoring and Remediation Training for Schizophrenia
Brief Title: Examining Strategy Monitoring and Remediation Training
Acronym: E-SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Michael Best, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 39698
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Psychotic Disorders; Executive Dysfunction
Keywords: psychosis; schizophrenia; cognitive remediation; executive functioning; strategy monitoring; computerized practice; cognitive training
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive Computerized Cognitive Training only, Strategy Development only, or both (Executive Functioning Training; ET).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be informed that they will be randomized to one of three types of cognitive training, however, will have no idea what the conditions or the hypotheses. Outcome assessors will be blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Executive Training (Active Comparator): The Executive Training (ET) condition will consist of the ET intervention that Dr. Best previously developed and evaluated. ET sessions consist of 50% of the session practicing computerized cognitive training exercises, and 50% of the session developing cognitive strategies to use in the computerized exercises. Participants are encouraged to complete 40 minutes of computerized training per day, and complete strategy worksheets, at home between sessions. All interventions will be delivered virtually in the participant's home and group sessions will be conducted using the online platform Zoom.
  Interventions: Other: Strategy Development; Other: Computerized Cognitive Training
- Strategy Development only (Experimental): In Strategy Development only participants will engage in cognitive strategy discussions to develop new executive function strategies that can be used in daily life. Between sessions, participants will be encouraged to practice their cognitive strategies in their daily life and track their strategies using the strategy worksheet. There will be no computerized cognitive training in this condition. All interventions will be delivered virtually in the participant's home and group sessions will be conducted using the online platform Zoom.
  Interventions: Other: Strategy Development
- Computerized Cognitive Training only (Experimental): In Computerized Cognitive Training only participants will spend the entire one-hour session practicing computerized training exercises. Between sessions participants will be encouraged to practice the computerized exercises at home for 40 minutes per day. There will be no strategy development in this condition. All interventions will be delivered virtually in the participant's home and group sessions will be conducted using the online platform Zoom.
  Interventions: Other: Computerized Cognitive Training

INTERVENTIONS:
Other: Strategy Development — Participants engage in cognitive strategy discussions to develop new executive function strategies that can be used in daily life, and track their strategies between sessions. No computerized cognitive training.
  Arms: Executive Training; Strategy Development only
Other: Computerized Cognitive Training — Participants practice computerized training exercises targeting executive functioning skills, and complete computerized exercises between sessions.
  Arms: Computerized Cognitive Training only; Executive Training

SUMMARY:
Executive Function Training is a cognitive training approach that specifically trains executive functioning for people with schizophrenia-spectrum disorders. The current study compares full executive function training to computerized training alone and to strategy monitoring alone.

DETAILED DESCRIPTION:
All interventions will involve 4 weeks of group treatment consisting of two 1-hour group sessions per week and additional practice at home between sessions. The Executive Training condition will consist of 50% of the session practicing computerized cognitive training exercises, and 50% of the session developing cognitive strategies to use in the computerized exercises. Participants are encouraged to complete 40 minutes of computerized training per day, and complete strategy worksheets, at home between sessions. In Computerized Cognitive Training only participants will spend the entire one-hour session practicing computerized training exercises. Between sessions participants will be encouraged to practice the computerized exercises at home for 40 minutes per day. There will be no strategy development in this condition. In Strategy Development only participants will engage in cognitive strategy discussions to develop new executive function strategies that can be used in daily life. Between sessions, participants will be encouraged to practice their cognitive strategies in their daily life and track their strategies using the strategy worksheet. There will be no computerized cognitive training in this condition. All interventions will be delivered virtually in the participant's home and group sessions will be conducted using the online platform Zoom.

90 participants with schizophrenia-spectrum disorders will be recruited. Power analyses, conducted with GPower, indicate that 90 participants (30 per treatment condition), accounting for an upper limit of 25% attrition observed in my previous trials of ET, provides 80% power to detect a medium effect size (cohen's f = 0.2) difference between conditions.

Primary and secondary outcomes will be examined using Linear Mixed Models on the Intent-to-Treat sample with missing data interpolated using maximum likelihood estimation. The primary endpoint is the 3-month follow-up assessment, and secondary endpoint of post-treatment will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of schizophrenia, schizoaffective disorder or any other psychotic disorder (based on DSM-V)
* 18-65 years of age
* know how to use a computer
* not abusing drugs or alcohol
* can read and speak English.

Exclusion Criteria:

* enrolled in a cognitive training program in the last 6 months
* neurological disease or neurological damage
* medical illnesses that can change neurocognitive function
* medical history of head injury with loss of consciousness
* physical handicaps

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Specific Levels of Functioning Scale | Change from Baseline to 12-Week Follow-up
  The SLOF is a behavioral questionnaire assessing community functioning. It includes 43 items, grouped into six subscales: Physical functioning; Personal care skills; Interpersonal relationships; Social acceptability; Activities of community living; and Work skills. Each of the 43 questions in the above subscales is rated on a 5-point Likert scale (1 = poorest function, 5 = best function) with anchors describing the frequency of the behavior and/or patient's level of independence. The higher the total score, the better the overall functioning of the individual. Scores range from 43 - 215.

SECONDARY OUTCOMES:
Cambridge Neuropsychological Test Automated Battery (CANTAB) | Change from Baseline to 12-Week Follow-up
  The CANTAB is a battery consisting of highly sensitive, precise and objective measures of cognitive function. It includes tests of working memory, learning and executive function; visual, verbal and episodic memory; attention, information processing and reaction time; social and emotion recognition, decision making and response control. A higher total score is indicative of better cognitive performance.
Wide Range Achievement Test (WRAT) | Change from Baseline to 12-Week Follow-up
  The WRAT is an academic skills assessment which measures reading skills, math skills, spelling, and comprehension. The WRAT-3 Reading is a letter and word recognition subtest assessing reading ability. It contains 15 letters and 42 words. The lowest possible score would be a 0 and the highest score would be a 57. Higher scores are indicative of better reading ability.
Questionnaire About the Process of Recovery (QPR) | Change from Baseline to 12-Week Follow-up
  The QPR was developed from service users' accounts of recovery from psychosis in collaboration with local service users. It asks people living with psychosis about aspects of recovery that are meaningful to them, and is strongly associated with general psychological wellbeing, quality of life and empowerment. There are 15 items rated from 0-4, so the minimum score is 0 and the maximum is 60. A higher score is indicative of greater personal recovery.
Brief Psychiatric Rating Scale (BPRS) | Change from Baseline to 12-Week Follow-up
  The BPRS is an assessor-rated and interview-based measure assessing psychopathology and symptom severity. There are 24 items rated from 1-7, with 1 representing "absent" and 7 representing "extremely severe". The minimum score is 24 and the maximum is 168. Higher scores are indicative of increased symptomology.
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | Change from Baseline to 12-Week Follow-up
  The Q-LES-Q is a 93-item self-report measure assessing the degree of enjoyment and satisfaction experienced in areas of daily functioning, including physical health/activities (13 items), feelings (14 items), work (13 items), household duties (10 items), school/course work (10 items), leisure time activities (6 items), social relations (11 items), and general activities (16 items). Responses are rated on a 5-point scale, with 1 being "not at all or never" or "very poor" and 5 being "frequently or all of the time" or "very good". The raw total score ranges from 93 to 465, with higher scores indicative of more enjoyment and satisfaction.
Dysfunctional Attitudes Scale (DAS) | Change from Baseline to 12-Week Follow-up
  DAS is a 40-item self-report measure assessing dysfunctional beliefs. The degree of agreement to each statement is scored on a 7-point Likert scale (1 = agree totally, 2 = agree very much, 3 = agree slightly, 4 = neutral, 5 = disagree slightly, 6 = disagree very much, 7 = disagree totally). The lowest possible scale is 40 while the highest possible scale is 280. Higher scores would indicate more negative beliefs.
Brief Core Schema Scale (BCSS) | Change from Baseline to 12-Week Follow-up
  The BCSS assesses four dimensions of self and other evaluation: negative-self, positive-self, negative-other, and positive-other. The BCSS have 24 items concerning beliefs about the self and others that are assessed on a ﬁve-point rating scale (0-4). Four scores are obtained: negative-self (six items), positive-self (six items), negative-others (six items) and positive-others (six items). Higher scores are indicative of stronger belief. Scores range from 0 - 96.
Generalized Self-Efficacy Scale (GSES) | Change from Baseline to 12-Week Follow-up
  The GSES assesses optimistic self-beliefs to cope with a variety of difficult demands in life. There are 10 items rated from 1-4, with 1 being "not at all true" and 4 being "exactly true". The lowest score possible is 10 and the highest is 40, with higher scores representing higher levels of optimistic self-beliefs.
Cognitive Failures Questionnaire (CFQ) | Change from Baseline to 12-Week Follow-up
  The CFQ is a 25-item self-report measure designed to assess perception, memory, and motor lapses in daily life. Frequency of experiencing each item is assessed on a 5-point scale, ranging from "0 = Never" to "4 = Very Often". The lowest score would be a 0 and the highest score would be a 100. Higher scores indicate more cognitive failures.
Need for Cognition Scale (NCS) | Change from Baseline to 12-Week Follow-up
  The NCS measures individual's tendency to engage in and enjoy thinking. Responses are rated on a 5-point scale, ranging from "1 = Extremely Unlike Me" to "5 = Extremely Like Me". The lowest score would be an 18 and the highest score would be a 90, with reverse scoring counted. Higher scores indicate increased tendency to engage in and enjoy thinking.
Davos Assessment of Cognitive Biases (DACOBS) | Change from Baseline to 12-Week Follow-up
  The DAVOS measures cognitive biases and discriminates between schizophrenia spectrum patients and normal control subjects. 42 items are scored from 1-7, with total scores ranging from 42-294. Higher scores indicate stronger beliefs/attitudes.
Motivation and Pleasure Scale - Self-Report (MAP-SR) | Change from Baseline to 12-Week Follow-up
  The MAP-SR is a 15-item self-report measure assessing the motivation and pleasure a person has experienced. (1) Social pleasure, (2) recreational or work pleasure, (3) feelings and motivations about close, caring relationships and (4) motivation and effort to engage in activities are evaluated. Responses are rated on a 5-point scale, where 0 represents "no pleasure", "not at all important to me", "not at all motivated", or "no effort", and 4 represents "extreme pleasure", "extremely important to me", "very motivated" or "very much effort". The highest score would be a 60 while the lowest score would be a 0. Higher scores indicate more pleasure and motivations.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Best, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto Scarborough, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu EQ, Birnbaum HG, Shi L, Ball DE, Kessler RC, Moulis M, Aggarwal J. The economic burden of schizophrenia in the United States in 2002. J Clin Psychiatry. 2005 Sep;66(9):1122-9. doi: 10.4088/jcp.v66n0906. PMID 16187769
- [Background] Palmer BA, Pankratz VS, Bostwick JM. The lifetime risk of suicide in schizophrenia: a reexamination. Arch Gen Psychiatry. 2005 Mar;62(3):247-53. doi: 10.1001/archpsyc.62.3.247. PMID 15753237
- [Background] Eack SM, Newhill CE. Psychiatric symptoms and quality of life in schizophrenia: a meta-analysis. Schizophr Bull. 2007 Sep;33(5):1225-37. doi: 10.1093/schbul/sbl071. Epub 2007 Jan 4. PMID 17204532
- [Background] Swartz MS, Perkins DO, Stroup TS, Davis SM, Capuano G, Rosenheck RA, Reimherr F, McGee MF, Keefe RS, McEvoy JP, Hsiao JK, Lieberman JA; CATIE Investigators. Effects of antipsychotic medications on psychosocial functioning in patients with chronic schizophrenia: findings from the NIMH CATIE study. Am J Psychiatry. 2007 Mar;164(3):428-36. doi: 10.1176/ajp.2007.164.3.428. PMID 17329467
- [Background] Eack SM, Hogarty GE, Cho RY, Prasad KM, Greenwald DP, Hogarty SS, Keshavan MS. Neuroprotective effects of cognitive enhancement therapy against gray matter loss in early schizophrenia: results from a 2-year randomized controlled trial. Arch Gen Psychiatry. 2010 Jul;67(7):674-82. doi: 10.1001/archgenpsychiatry.2010.63. Epub 2010 May 3. PMID 20439824
- [Background] Subramaniam K, Luks TL, Fisher M, Simpson GV, Nagarajan S, Vinogradov S. Computerized cognitive training restores neural activity within the reality monitoring network in schizophrenia. Neuron. 2012 Feb 23;73(4):842-53. doi: 10.1016/j.neuron.2011.12.024. PMID 22365555
- [Background] Best MW, Milanovic M, Iftene F, Bowie CR. A Randomized Controlled Trial of Executive Functioning Training Compared With Perceptual Training for Schizophrenia Spectrum Disorders: Effects on Neurophysiology, Neurocognition, and Functioning. Am J Psychiatry. 2019 Apr 1;176(4):297-306. doi: 10.1176/appi.ajp.2018.18070849. Epub 2019 Mar 8. PMID 30845819
- [Background] Best MW, Gale D, Tran T, Haque MK, Bowie CR. Brief executive function training for individuals with severe mental illness: Effects on EEG synchronization and executive functioning. Schizophr Res. 2019 Jan;203:32-40. doi: 10.1016/j.schres.2017.08.052. Epub 2017 Sep 19. PMID 28931460
- [Background] Wykes T, Spaulding WD. Thinking about the future cognitive remediation therapy--what works and could we do better? Schizophr Bull. 2011 Sep;37 Suppl 2(Suppl 2):S80-90. doi: 10.1093/schbul/sbr064. PMID 21860051
- [Background] Best MW, Bowie CR. A review of cognitive remediation approaches for schizophrenia: from top-down to bottom-up, brain training to psychotherapy. Expert Rev Neurother. 2017 Jul;17(7):713-723. doi: 10.1080/14737175.2017.1331128. Epub 2017 May 24. PMID 28511562
- [Background] Ruse SA, Harvey PD, Davis VG, Atkins AS, Fox KH, Keefe RS. Virtual Reality Functional Capacity Assessment In Schizophrenia: Preliminary Data Regarding Feasibility and Correlations with Cognitive and Functional Capacity Performance. Schizophr Res Cogn. 2014 Mar;1(1):e21-e26. doi: 10.1016/j.scog.2014.01.004. PMID 25083416
- [Background] Neil ST, Kilbride M, Pitt L, Nothard S, Welford M, Sellwood W, Morrison AP. The questionnaire about the process of recovery (QPR): A measurement tool developed in collaboration with service users. Psychosis. 2009; 1(2): 145-155.
- [Background] Faustman WO, Overall JE. (1999). Brief Psychiatric Rating Scale. In M. E. Maruish (Ed.), The use of psychological testing for treatment planning and outcomes assessment (p. 791-830). Lawrence Erlbaum Associates Publishers.
- [Background] Endicott J, Nee J, Harrison W, Blumenthal R. Quality of Life Enjoyment and Satisfaction Questionnaire: a new measure. Psychopharmacol Bull. 1993;29(2):321-6. PMID 8290681
- [Background] Weissman AN, Beck AT. Development and validation of the dysfunctional Attitude Scale: A preliminary investigation. Paper presented at the Association for the Advancement of Behavior Therapy; Chicago. 1978.
- [Background] Fowler D, Freeman D, Smith B, Kuipers E, Bebbington P, Bashforth H, Coker S, Hodgekins J, Gracie A, Dunn G, Garety P. The Brief Core Schema Scales (BCSS): psychometric properties and associations with paranoia and grandiosity in non-clinical and psychosis samples. Psychol Med. 2006 Jun;36(6):749-59. doi: 10.1017/S0033291706007355. Epub 2006 Mar 27. PMID 16563204
- [Background] Schwarzer R, Jerusalem M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, UK: NFER-NELSON.
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Cacioppo JT, Petty RE, Quintanar LR. Individual differences in relative hemispheric alpha abundance and cognitive responses to persuasive communications. J Pers Soc Psychol. 1982 Sep;43(3):623-36. doi: 10.1037//0022-3514.43.3.623. PMID 7131245
- [Background] van der Gaag M, Schutz C, Ten Napel A, Landa Y, Delespaul P, Bak M, Tschacher W, de Hert M. Development of the Davos assessment of cognitive biases scale (DACOBS). Schizophr Res. 2013 Mar;144(1-3):63-71. doi: 10.1016/j.schres.2012.12.010. Epub 2013 Jan 15. PMID 23332365
- [Background] Llerena K, Park SG, McCarthy JM, Couture SM, Bennett ME, Blanchard JJ. The Motivation and Pleasure Scale-Self-Report (MAP-SR): reliability and validity of a self-report measure of negative symptoms. Compr Psychiatry. 2013 Jul;54(5):568-74. doi: 10.1016/j.comppsych.2012.12.001. Epub 2013 Jan 22. PMID 23351831
- See also: CANTAB Virtual Assessment — http://www.cantab.com
- See also: WRAT-5: Wide Range Achievement Test Professional Manual — https://books.google.ca/books?id=amQXtAEACAAJ

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT04756388/Prot_SAP_000.pdf